CLINICAL TRIAL: NCT01574729
Title: Phase II Study of Surgery Combined With Recombinant Adenoviral Human p53 Gene Therapy in Treatment Advanced Non-small-cell Carcinoma
Brief Title: Surgery Combined With rAd-p53 Gene in Treatment Advanced Non-small-cell Carcinoma
Acronym: rAd-p53
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shenzhen SiBiono GeneTech Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: rAd-p53NSCLC
Record Dates: First submitted 2012-04-06; First posted 2012-04-10 (Estimated); Last update posted 2012-06-28 (Estimated); Status verified 2012-06

CONDITIONS: Non-small Cell Lung Cancer
Keywords: p53 gene therapy; non-small cell lung cancer; post-surgery; chemotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Surgery plus post-surgery chemotherapy (Active Comparator): Surgery plus post-surgery chemotherapy
  Interventions: Procedure: Surgery
- Surgery combined with rAd-p53 gene therapy (Experimental): Surgery combined with the surgery wound surface injection of rAd-p53 plus post-surgery chemotherapy
  Interventions: Drug: Surgery combined with rAd-p53 gene therapy

INTERVENTIONS:
Drug: Surgery combined with rAd-p53 gene therapy — Surgery combined with rAd-p53 gene therapy during surgery plus post-surgery chemotherapy
  Arms: Surgery combined with rAd-p53 gene therapy
Procedure: Surgery — Surgery plus post-surgery chemotherapy
  Arms: Surgery plus post-surgery chemotherapy

SUMMARY:
The primary objectives of this study are to investigate the efficacy and safety of surgery combined with rAd-p53 gene therapy in treatment of advanced Non-small-cell lung carcinoma (NSCLC). The study efficacy endpoints include overall survival, progress-free survival, quality of life, and local recurrent rate. The safety endpoint is complications and adverse effects.

The study hypothesis: rAd-p53 gene therapy can prolong the overall survival and reduce the local recurrent rate.

ELIGIBILITY:
Inclusion Criteria:

* historically diagnosed advanced non-small lung cancer
* has surgery indication
* age 18 years old or greater
* life expectancy greater than 12 weeks
* ECOG: 0-2
* no prior chemotherapy, radiotherapy in 2 weeks
* Neutrophils≥1.5×10^9/L,platelet≥80×10^9/L, Hb≥≥80g/L,bilirubin≤1.5×2mg/dl, ALT and AST≤2×institutional upper limit of normal,Cr≤1.5×institutional upper limit of normal,coagulation tests(INR and PTT)within normal range
* subject provides signed informed consent

Exclusion Criteria:

* hypersensitive to study drug
* with a coagulational test unnormal or a bleeding disorder
* infections
* with serious condition which can't stand a surgery
* pregnant or lactating
* principle investigator consider not suitable

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2012-08; Primary Completion 2015-08 (Estimated); Study Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
overall survival | 3 year after the treatment
  determine the 3-years overall survival
adverse effects | from starting treatment to 30 days after treatment

SECONDARY OUTCOMES:
local recurrent rate | 3 years
quality of life | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Qunyou Tan, M.D., Ph.D, Principal Investigator — Institute of Surgery Research, Daping Hospital, Third Military Medical University
Locations (1):
- Institute of Surgery Research, Daping Hospital, Third Military Medical University, Chongqing, Chongqing Municipality, China